CLINICAL TRIAL: NCT02825758
Title: A Study to Evaluate the Acceptability of ZestiVits; a New Vitamin, Mineral and Trace Element Supplement for Those Aged 11 and Over on a Ketogenic or Restricted Diet With Regard to Product Tolerance, Palatability and Compliance
Brief Title: Evaluation of ZestiVits in Children and Adults on a Ketogenic or Restricted Therapeutic Diet
Acronym: ZestiVits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vitaflo International, Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCT-Zest-14/01/2016-01; 209722 (Other: IRAS)
Record Dates: First submitted 2016-06-24; First posted 2016-07-07 (Estimated); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Deficiency of Micronutrients
Keywords: Micronutrients; restricted; ketogenic; diet; acceptability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ZestiVits (Experimental): Supplement for use in ketogenic and restricted therapeutic diets, from the age of 11.
  Daily use for 7 days. Daily intake level for each subject will be determined and prescribed by a dietitian.
  Interventions: Dietary Supplement: ZestiVits

INTERVENTIONS:
Dietary Supplement: ZestiVits — The study product is a low-carbohydrate, orange flavour, vitamin, mineral and trace element (micronutrient) supplement for use in ketogenic and restricted therapeutic diets, for children aged from 11 years of age and adults.
  The recommended dosage of the study product for each subject will be determined and prescribed by a dietitian. This will be based on individual requirements for micronutrient supplementation.

SUMMARY:
A study to evaluate the acceptability of ZestiVits; a new vitamin, mineral and trace element supplement for children aged 11 years and over and adults on a ketogenic or restricted therapeutic diet with regard to product tolerance, palatability and compliance.

DETAILED DESCRIPTION:
To evaluate the gastrointestinal tolerance, palatability and compliance of ZestiVits in a seven-day period for 15 subjects aged 11 years and over following a ketogenic or restricted therapeutic diet.

* Qualitative assessments from subject questionnaires that allow evaluation of the acceptability and ease of use of the study product.
* Collection of daily data about the gastro-intestinal tolerance of the study product.

  * Collection of daily data about compliance with the study product i.e. actual versus prescribed intake.
  * Improve quality of life by increasing range of products available for use in a ketogenic or restricted therapeutic diet.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of condition requiring a ketogenic or restrictive therapeutic diet
2. On a ketogenic or restricted therapeutic diet with good compliance
3. Aged 11 years and over
4. Has a requirement for a micronutrient supplement
5. Written informed consent by subject or parent/carer

Exclusion Criteria:

1. Participants aged less than 11 years
2. Use of additional micronutrient supplements during the study period unless clinically indicated and prescribed by the investigator (must be recorded in patient case record file)

Min Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Palatability via qualitative assessments from a subject questionnaire | 7 days
  Qualitative outcome measures will be described in a narrative summarising the study outcomes
Gastrointestinal tolerance via qualitative assessments from a subject questionnaire | 7 days
  Qualitative outcome measures will be described in a narrative summarising the study outcomes
Patient compliance via qualitative assessments from a subject questionnaire | 7 days
  Qualitative outcome measures will be described in a narrative summarising the study outcomes
Ease of use of product via qualitative assessments from a subject questionnaire | 7 days
  Qualitative outcome measures will be described in a narrative summarising the study outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Gisela Wilcox, Principal Investigator — Northern Care Alliance NHS Foundation Trust
Locations (3):
- United Kingdom (3):
  - Bristol Royal Hospital for Children, Bristol, Avon
  - Salford Royal NHS Foundation Trust, Salford, Greater Manchester
  - Leeds Children's Hospital, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: No